CLINICAL TRIAL: NCT02552095
Title: A Prospective, Single Arm, Multi Center Study on the Compatibility of Triathlon PKR and the Motion Analysis for Japanese
Brief Title: Triathlon PKR Study in Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJCR-OR-1302
Record Dates: First submitted 2015-08-10; First posted 2015-09-16 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon PKR (Other): Patient who receives the Triathlon.
  Interventions: Device: Triathlon PKR

INTERVENTIONS:
Device: Triathlon PKR

SUMMARY:
The Purpose of this study is to evaluate compatibility of the Triathlon Partial Knee Replacement (PKR) with the Japanese population. It is expected that patients who receive the Triathlon PKR will achieve excellent clinical results without adverse effects and that the device fits well with Japanese morphology.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requires a primary unicompartmental knee replacement.
2. Patient is between 20 years old to 80 years old.
3. Patient is diagnosed as osteoarthritis, rheumatoid arthritis, traumatic arthritis or avascular necrosis.
4. Patient can walk independently at least 10m.
5. Patient has signed the Institutional Review Board (IRB) approved, study specific informed patient consent form.
6. Patient is willing and able to comply with post-operative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient requires a revision.
2. Patient is pregnant.
3. Patient has lateral osteoarthritis.
4. Patient has less than 10°of flexion contracture and greater than 90°of flexion.
5. Patient's preoperative mechanical alignment is less than 10° of varus and 15° of valgus.
6. Patient has had high tibial osteotomy, femoral osteotomy and/or joint fusion.
7. Patient has a neuromuscular or neurosensory deficiency that would limit the ability to assess the performance of the device.
8. Patient has a systemic or metabolic disorder leading to progressive bone deterioration.
9. Patient is immunologically suppressed or receiving steroids (>30 days) in excess of normal physiological requirements.
10. Patient has a deformity which will require the use of wedges or augments.
11. Patient has an active or suspected latent infection in or about the knee joint.
12. Patient who is inappropriate for participating in the study by the judgment of the investigator.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-operation, 6 months, 12 months and 24 months after surgery

SECONDARY OUTCOMES:
Measurement of tibial resection plane (A-P length and width of resection) | intraoperative
Change in Quality of life as assessed by 12-Item Short-Form Health Survey (SF-12) questionnaire | Pre-operation, 6 months, 12 months and 24 months after surgery
Change in Japanese Orthopaedics Association (JOA) score | Pre-operation, 6 months, 12 months and 24 months after surgery

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Kushiro-sanjikai Hospital, Kushiro, Hokkaido
  - Akabane Central General Hospital, Tokyo, Kita-ku
  - Toneyama National Hospital, Toyonaka, Osaka
  - Nihon University Hospital, Itabashi-ku, Tokyo
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto